CLINICAL TRIAL: NCT06755021
Title: Whey Protein Milk-Derived Exosomes Among Ulcerative Colitis Patients
Brief Title: Whey Protein Milk-Derived Exosomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Exosomm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WPMDE2
Record Dates: First submitted 2024-12-11; First posted 2025-01-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: The interventional group will be divided into two sub-groups for supplement dosage.
  Group 1 will receive 5g of WPMDE twice daily, while Group 2 will receive 10g of WPMDE twice daily.
Masking Description: open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with ulcerative colitis (UC) of varying disease severity, ranging from mild to severe (Experimental): Participants will be sequentially allocated to the two dosage groups in a 1:1 ratio: dosage X and dosage 2X and stratified by disease severity
  Interventions: Dietary Supplement: Whey Protein Milk-Derived Exosomes

INTERVENTIONS:
Dietary Supplement: Whey Protein Milk-Derived Exosomes — WPMDE2 (Whey Protein Milk-Derived Exosomes 2) is an advanced nutritional supplement developed from natural milk components.

SUMMARY:
This Phase 1B open-label, uncontrolled multicenter trial evaluates the safety, tolerability, and potential efficacy of WPMDE2, a whey protein milk-derived exosome supplement, in adult patients with mild to severe ulcerative colitis (UC). The study aims to explore clinical improvements in disease activity, quality of life, and inflammatory markers over an 8-week intervention period with a 2-week follow-up. WPMDE2 is administered orally in two dosage groups, with 100 participants stratified by disease severity. Key endpoints include changes in disease severity, fecal calprotectin levels, and patient-reported outcomes. Conducted under ethical guidelines, the study seeks to establish WPMDE2 as a safe, naturally derived adjunct therapy for UC patients.

DETAILED DESCRIPTION:
This is a Phase 1B open-label, uncontrolled, multicenter trial designed to evaluate the safety, tolerability, and potential efficacy of WPMDE2 (Whey Protein Milk-Derived Exosomes) in adult patients with varying severities of ulcerative colitis (UC). The study builds upon promising preclinical research and a preceding Phase 1 safety study in healthy volunteers, which demonstrated that WPMDE2 has a favorable safety profile and potential anti-inflammatory benefits. By targeting patients with mild to severe UC, the trial seeks to explore WPMDE2's therapeutic role as an add-on to existing treatment regimens.

Study Objectives

Primary Objectives:

Evaluate the safety and tolerability of WPMDE2 when administered orally at two different dosages.

Assess the clinical benefits of WPMDE2 by measuring changes in disease severity.

Secondary Objectives:

Investigate improvements in quality of life (QoL) using the IBDQ-32 questionnaire.

Monitor changes in inflammatory biomarkers, including fecal calprotectin. Assess endoscopic improvements and other patient-reported outcomes, such as stool frequency, rectal bleeding, and abdominal pain.

Study Design This trial is an open-label, uncontrolled study involving multiple centers in Israel, with potential sites abroad. Participants will receive WPMDE2 in one of two dosage groups (X and 2X) for 8 weeks, followed by a 2-week follow-up period. The design accommodates real-world applicability by allowing participants to continue their standard UC treatments while taking WPMDE2.

Key Features:

Study Type: Interventional Intervention Model: Sequential allocation into two dosage groups. Primary Purpose: Exploratory evaluation of safety and efficacy. sample size:

A total of 100 patients with confirmed UC will be enrolled:

Intervention Details

Product Description:

WPMDE2 is a powder derived from milk, enriched with naturally occurring extracellular vesicles (EVs). These EVs contain bioactive components, including proteins, lipids, and microRNAs, which exhibit immunomodulatory and anti-inflammatory properties. Participants will take the powder dissolved in water twice daily, with doses stratified into two groups: 5g and 10g.

WPMDE2 has been optimized to preserve the structural integrity of its active components. Its safety was confirmed in Phase 1 studies involving healthy volunteers.

Administration:

Participants will be provided with pack with powder with measuring spoon to prepare the solution.Oral administration will occur twice daily for 8 weeks.

Study Procedures

Participants will attend four scheduled visits:

V0 (Screening): Initial assessment, including blood and stool tests, endoscopic evaluation (optional), and eligibility screening.

V1 (Baseline): Randomization and initial intervention. V2 (End of Treatment): Final assessment of treatment impact, including blood and stool tests, endoscopic evaluation, and patient-reported outcomes.

V3 (Follow-up): Virtual visit 2 weeks post-treatment for safety monitoring. Daily Diaries: Participants will record adherence, symptoms (e.g., rectal bleeding, stool frequency), and any new medications.

*Colonoscopy will be considered the gold standard for the diagnosis of ulcerative colitis (UC). Before recruitment, colonoscopy results will be collected for each subject to evaluate and determine the diagnosis of UC. Only available examination results that meet the study's needs will be collected.

At the end of the trial (EOT), a colonoscopy will be performed based on the sponsor's decision, with a maximum of 15 subjects eligible. Participation in this examination will be optional.

For patients who consent to endoscopic evaluation, special attention will be given to the quality control of endoscopic data. A central reviewer will assess all endoscopic images to ensure consistent scoring across sites. However, since endoscopy is optional, the analysis plans will account for potential missing endoscopic data.

Endpoints

Primary Endpoints:

Changes in disease severity from baseline to week 8. Incidence of adverse events and changes in vital signs or laboratory results.

Secondary Endpoints:

Reduction in inflammatory biomarkers, such as fecal calprotectin. Endoscopic improvement in mucosal healing. Improvements in quality of life as measured by IBDQ-32. Patient-reported outcomes, including stool frequency and abdominal pain. Statistical Considerations Sample Size: 100 participants, providing sufficient power to detect meaningful differences.

Analysis Populations: Intention-to-Treat (ITT) and Per-Protocol (PP).

Handling Missing Data: Multiple imputation techniques will ensure robust ITT analysis.

Ethical Considerations The study adheres to the Declaration of Helsinki and relevant regulatory guidelines. Ethical approval has been obtained from IRBs at participating centers. Participants will provide informed consent before enrolling, and their safety will be closely monitored throughout the study. Adverse events will be reported promptly, with provisions for discontinuing the intervention if necessary.

Expected Outcomes If successful, this trial will provide evidence for WPMDE2 as a safe, naturally derived adjunct therapy for UC. Findings will inform the design of future controlled trials, potentially leading to a novel therapeutic option for patients with inflammatory bowel disease.

Timelines Site Initiation: Within 3 month of IRB approval. Recruitment: Over 8 months. Intervention Period: 8 weeks per participant. Follow-up and Analysis: Completed within 3 months of the last patient visit. This study represents an innovative approach to leveraging milk-derived bioactive components to address unmet needs in UC management.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed clinical diagnosis of UC of any duration
* Age 18-65 years
* Signed informed consent
* Presence of endoscopic evidence of colonic inflammation

Exclusion Criteria:

* Pregnancy or breastfeeding
* Milk allergy
* Severe co-morbid medical illness such as uncontrolled diabetes, unstable cardiovascular or pulmonary disease, or malignancy
* Specific exclusions: HIV , CMV , Hepatitis B or C, Abnormal AST or ALT at screening defined as > 3x upper limit of normal
* Participating in another investigational drug study within 30 days of study enrollment
* Evidence of colonic perforation
* Massive hemorrhage from the colon requiring emergent surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit #1 | 12 months
  - Change in disease activity as measured by clinical activity index from baseline to end of treatment
Clinical Benefits #2 | 12 months
  - Comparison of clinical benefits between the two dosage groups measured by clinical activity index from baseline to end of treatment
Safety and Tolerability of WPMDE2 #1 | 12 months
  - Incidence and severity of adverse events.

SECONDARY OUTCOMES:
Change in inflammatory biomarkers #1 | 12 months
  - Fecal calprotectin levels
Change in inflammatory biomarkers #2 | 12 months
  - Change in endoscopic subscore of the clinical activity index from baseline to end of treatment
Improvement in the quality of life | 12 months
  Improvement in the quality of life as measured by IBDQ-32
Patient-reported outcomes #1 | 12 months
  Changes in stool frequency assessed by the IBDQ-32 questionnaire Changes in rectal bleeding Changes in abdominal pain/discomfort
Patient-reported outcomes #2 | 12 months
  Changes in rectal bleeding assessed by the IBDQ-32 questionnaire
Dose-response relationship: | 12 months
  Comparison of all endpoints between the two dosage groups to assess dose-response effects measured by the change in clinical activity index from baseline to end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Kats, MD, Principal Investigator — Hadassah Medical Organization